CLINICAL TRIAL: NCT07400770
Title: Effect of a Snyder Hope Theory-Based Nursing Intervention on Psychological Status, Pain, and Functional Recovery in Elderly Patients After Hip Fracture Surgery: A Randomized Controlled Trial
Brief Title: Hope Theory-Based Nursing Intervention After Hip Fracture Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Orthopaedic Surgery, Taizhou No.3 People's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TZSRY-HIP-HOPE-2024
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hip Fracture; Elderly Patients; Postoperative Recovery; Nursing Interventions; Snyder Hope Theory
Keywords: Hope Theory; Elderly Hip Fracture Surgery; Postoperative Nursing; Psychological Counseling; Rehabilitation Training; Pain Management, Anxiety; Quality of Life
MeSH Terms: conditions — Hip Fractures; Agnosia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial with two parallel groups: an experimental group receiving Snyder Hope Theory-based nursing intervention and a control group receiving standard postoperative care. The intervention involves psychological counseling, goal-setting, rehabilitation training, and peer support. The effectiveness of the intervention will be measured using Herth Hope Index, Visual Analog Scale for pain, Harris Hip Score for hip joint function, and WHOQOL-BREF for quality of life assessment.
Masking Description: This is an open-label study, meaning there is no masking for the participants, care providers, investigators, or outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snyder Hope Theory-based Nursing Intervention (Experimental): Participants in the intervention arm will receive a Snyder Hope Theory-based nursing intervention, which includes psychological counseling, goal-setting, rehabilitation training, and peer support to improve hope levels, reduce pain, and enhance functional recovery after hip fracture surgery.
  Interventions: Behavioral: Snyder Hope Theory-based Nursing Intervention
- Standard Postoperative Care (Active Comparator): Participants in the control arm will receive standard postoperative care, including routine pain management, rehabilitation exercises, and general guidance on recovery after hip fracture surgery, without the addition of the Snyder Hope Theory-based intervention.
  Interventions: Behavioral: Standard Postoperative Care

INTERVENTIONS:
Behavioral: Snyder Hope Theory-based Nursing Intervention — The Snyder Hope Theory-based nursing intervention involves a structured program aimed at improving the psychological well-being and recovery of elderly patients post-hip fracture surgery. The intervention includes psychological counseling, rehabilitation goal-setting, peer support, and motivation enhancement. The nursing intervention is designed to increase hope levels, reduce pain, alleviate anxiety, and improve hip joint function, ultimately enhancing the overall recovery process for the participants.
  Arms: Snyder Hope Theory-based Nursing Intervention
Behavioral: Standard Postoperative Care — Participants in the control group will receive standard postoperative care, including routine pain management, rehabilitation exercises, and general guidance on recovery after hip fracture surgery, without the addition of the Snyder Hope Theory-based intervention.
  Arms: Standard Postoperative Care

SUMMARY:
This is a randomized controlled trial to evaluate the effectiveness of a Snyder Hope Theory-based nursing intervention on elderly patients following hip fracture surgery. The study aims to improve the patient's psychological well-being, reduce pain, and enhance their functional recovery. Participants will be randomly assigned to either the intervention group or the control group. The intervention involves individualized counseling, goal setting, and rehabilitation training based on the Snyder Hope Theory. The trial will assess changes in hope levels, anxiety, pain, hip joint function, and quality of life before and after the intervention.

DETAILED DESCRIPTION:
This clinical trial aims to explore the impact of a Snyder Hope Theory-based nursing intervention on elderly patients who have undergone hip fracture surgery. As hip fractures are common among the elderly and often result in prolonged recovery periods, pain, and anxiety, effective interventions are needed to improve recovery outcomes.

In this study, elderly patients over the age of 60, who have undergone hip fracture surgery, will be recruited. They will be randomly assigned to either the intervention group or the control group. The intervention group will receive a specialized nursing care plan incorporating elements of the Snyder Hope Theory, including personalized psychological counseling, rehabilitation goal-setting, and group-based support. The control group will receive standard postoperative care.

The primary outcomes include the improvement in hope levels (measured by the Herth Hope Index), reduction in pain (measured by the Visual Analog Scale), and enhanced physical function (measured by the Harris Hip Score). Secondary outcomes include anxiety reduction and quality of life improvement (measured by the WHOQOL-BREF).

The trial will be conducted over a 2-week period, with assessments before and after the intervention. Data will be analyzed to determine the effectiveness of the intervention in improving psychological, functional, and physical outcomes for elderly patients recovering from hip surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years.
* Patients with hip fracture requiring surgical intervention.
* Patients who have undergone hip fracture surgery within the past 2 weeks.
* Patients who are able to communicate and provide informed consent.
* Patients and/or their family members who are willing to participate in the study.

Exclusion Criteria:

* Patients with other lower limb fractures or history of lower limb thrombosis.
* Patients with multiple fractures.
* Patients with severe damage to major organs (heart, lungs, brain) or malignant tumors.
* Patients who have undergone hip replacement surgery in the past.
* Patients with infectious diseases or immune system disorders.
* Patients with chronic diseases or neurological disorders.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Hope Levels (Herth Hope Index) | Pre-intervention and post-intervention (2 weeks)
  The primary outcome measure is the change in the patients' hope levels, which will be assessed using the Herth Hope Index. This scale is designed to measure the psychological and emotional dimensions of hope, focusing on the patients' expectations and their outlook on recovery and life. The Herth Hope Index will be administered before and after the intervention to assess changes in hope levels.

SECONDARY OUTCOMES:
Pain Level (VAS) | Pre-intervention and post-intervention (2 weeks)
  Pain levels will be assessed using the Visual Analog Scale (VAS), which measures the intensity of pain experienced by the patient on a scale from 0 (no pain) to 10 (worst possible pain). This measure will be used to evaluate the reduction of pain after the intervention.
Anxiety (STAI) | Pre-intervention and post-intervention (2 weeks)
  Anxiety levels will be assessed using the State-Trait Anxiety Inventory (STAI), a questionnaire that measures both state anxiety (temporary anxiety in a specific situation) and trait anxiety (general anxiety tendency). The tool will assess changes in anxiety after the intervention.
Hip Joint Function (Harris Hip Score) | Pre-intervention and post-intervention (2 weeks)
  Hip joint function will be assessed using the Harris Hip Score, which evaluates pain, function, and range of motion in the hip joint. This score helps in measuring functional recovery after hip fracture surgery.
Quality of Life (WHOQOL-BREF) | Pre-intervention and post-intervention (2 weeks)
  Quality of life will be measured using the WHOQOL-BREF, a brief version of the World Health Organization Quality of Life assessment. This tool evaluates physical health, psychological health, social relationships, and environment. It will assess improvements in the participants' overall quality of life post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Taizhou No. 3 People's Hospital, Taizhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No